CLINICAL TRIAL: NCT06080542
Title: Influence of Aerobic Exercise and HIIT on Glycemic Control in Adult Men With Type 1 Diabetes (TAILOR/1b)
Acronym: TAILOR/1b
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government); Ministerio de Ciencia e Innovación, Spain (Other Government); European Regional Development Fund (Other); Universitat Politècnica de València (Other)
Responsible Party: Principal Investigator, Rodrigo Martín-San-Agustin, Professor, University of Valencia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1587001
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: aerobic; men; glycemic; hiit
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Multiple Endocrine Neoplasia Type 1 | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Two interventions will be carried out in a single group, one aerobic session and HIIT session.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic session (Experimental): The aerobic exercise session will begin with a 3 min resting period (sitting quietly on the cycle ergometer (0 W), followed by a 3 min warm-up at 60 W and a stepwise intensity increase by 20 W / min (to control for day-to-day variations in exercise response) until the 5% of Pmax from IET above PLTP1 is achieved (i.e. moderate steady state walking or low-intensity running or cycling). This target workload will be maintained for 30 min. Active and passive recovery periods of 3 min each will be the same as the incremental test.
  Interventions: Procedure: Aerobic
- High-intensity interval training (Experimental): Our elastic band protocol is a modification of the HIIT protocols used by previous authors changing body weight exercises by exercises with TheraBand CLX. The exercise program is chosen to involve large muscle groups simulating conventional bodybuilding exercises by applying the external load to the elastic band's resistance. Four exercises of upper limb (bench press, seated dumbbell, shoulder press, and seated row) and four of lower limb (squats, stiff-legged deadlift, hamstring curl exercise, and quadriceps curl exercise) are chosen, which are intercalated in the program without doing two consecutive exercises of the same area. All exercises are done with both arms or legs at the same time.
  Interventions: Procedure: High-intensity interval training

INTERVENTIONS:
Procedure: Aerobic — This session will consist of an aerobic training session performed on a cycle ergometer.
  Arms: Aerobic session
Procedure: High-intensity interval training — This session will consist of a HIIT performed with elastic bands
  Arms: High-intensity interval training

SUMMARY:
Physical exercise is one of the main recommendations included in clinical guidelines for people with type 1 diabetes (T1D) because it is associated with substantially lower cardiovascular and overall mortality risks. Adherence to regular physical activity is low in the T1D population due to factors like time limitations, no access to appropriate equipment at home, or economic costs. High-intensity interval training (HIIT) has been proposed as a time-efficient methodology, consisting of sessions of short duration and high intensity exercises. An easier and cheaper training alternative for HIIT is exercising with elastic bands, either in a clinic or at home. Even so, training with elastic bands in T1D in combination with the HIIT method has not been compared to aerobic training. Besides, it is necessary to understand the glycemic impact of both kinds of exercise in order to build better artificial pancreas systems able to deal with exercise automatically. The aim of the study will be to determine the impact of aerobic exercise versus high-intensity interval training (HIIT) exercise on glycemic control.

DETAILED DESCRIPTION:
This HIIT modality presents differences with respect to other studies since it consists of strength exercises with elastic bands. This novelty represents an advantage because it can be an easier training alternative to perform in a clinical or home setting, compared to previous studies where cycle ergometer is used. Thus, one session of each type of exercise will be performed.

Prior to the exercise sessions, an incremental exercise test will be performed to determine the working power in the cycle ergometer. At the beginning of the test, subjects will be sit quietly on the cycle ergometer for 3 min (0 W) before they will start the warm-up period of 3 min with cycling at a workload of 60 W. Then, the workload will increase by 40 W every 3 min until volitional exhaustion. Finally, 3 min active recovery at 60 W followed by 3 min passive recovery (0 W) will be conducted on the cycle ergometer. Lactate turn point 1 (LTP1) and maximum power (Pmax) will be determined in order to prescribe the exercise intensity. Additionally, patients will conduct a familiarization session with the strength exercises in order to adapt the participants to exercises with elastic bands. Thus, the subjects will perform two sets of twelve repetitions of the exercises.

The aerobic exercise session will begin with a 3 min resting period (sitting quietly on the cycle ergometer (0 W), followed by a 3 min warm-up at 60 W and a stepwise intensity increase by 20 W / min (to control for day-to-day variations in exercise response) until the 5% of Pmax from IET above PLTP1 is achieved (i.e. moderate steady state walking or low-intensity running or cycling). This target workload will be maintained for 30 min. Active and passive recovery periods of 3 min each will be the same as the incremental test.

The elastic band protocol is a modification of the HIIT protocols used by previous authors changing body weight exercises by exercises with TheraBand CLX. The exercise program is chosen to involve large muscle groups simulating conventional bodybuilding exercises by applying the external load to the elastic band's resistance. Four exercises of upper limb (bench press, seated dumbbell, biceps curl, and seated row) and four of lower limb (squats, stiff-legged deadlift, hamstring curl exercise, and quadriceps curl exercise) are chosen, which are intercalated in the program without doing two consecutive exercises of the same area. All exercises are done with both arms or legs at the same time.

Prior to HIIT session, participants will carry out a warm-up consisting of 3 minutes at 60 W on the cycle ergometer and 15 no-load shoulder flexo-extensions. Session consists of two set of exercise intervals of 20s separated by 10s of rest (i.e. 4min in total) with a rest of 3 minutes between both series, making at each interval a different exercise resisted by the elastic band. The participants have to choose a width in the elastic band grip that supposed a maximum effort for the 20s of each exercise. Subjects will be encouraged to perform as many repetitions per interval as possible while maintaining correct form.

Perceived exertion will be used to determine the correct intensity of HIIT sessions. Immediately following each set of eight intervals, subjects will report ratings of perceived exertion using the Thera-Band resistance exercise scale of perceived exertion with Thera-Band® resistance bands. HIIT sessions correspond to a "Maximal". Heart rate will be measured continuously via chest belt telemetry (Polar H10) during all tests and also averaged over 5s.

A sample size of n=40 will be chosen for each study.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-40 years
* T1D with a diabetes duration for more than 2 years
* glycated hemoglobin (HbA1c) < 8.5% (<69 mmol mol-1)
* stable insulin regimen in the past 6 months with less than 20% change in total insulin daily dose
* multiple daily injections
* weekly physical activity of 90 min or more, but no practicing any sport as amateur or professional

Exclusion Criteria:

* clinical conditions or use of medications (other than insulin) known to affect glycemic control (e.g., oral/parenteral steroids or metformin, among others).

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Blood glucose Glucose control | The evaluated time points for exercise will be at 20 and 10 minutes before the session, at the beginning of the training and at 10, 20, and 30 minutes during the interval, and at 10 and 20 minutes after finishing the training.
  Blood glucose (mg/dL) will be measured through blood draws and YSI analysis
Interstitial glucose | 24 h pre-intervention and 24h post-intervention
  Interstitial glucose will be measured using the Dexcom G6 and FreeStyle 2 as a continuous glucose meters.
  Mean glucose, glycemic variability (measured using the Coefficient of Variation-CV) and the time spent at each glucose range [euglycemia (70-180 mg/dL) or Time in range (TIR), level 1 or mild hypoglycemia (54-70 mg/dL), level 2 or severe hypoglycemia (<54 mg/dL), level 1 hyperglycemia (180-250 mg/dL) and level 2 hyperglycemia (>250 mg/ dL)] will be evaluated with continuous glucose meters during 6 h, 12 h, and 24 h following both exercise sessions. Glucose before exercise were monitored using samples from a continuous glucose meters corresponding to a window of 24 hours before the exercise that exactly correspond to the clock times of the patient in the 24h after the exercise

SECONDARY OUTCOMES:
Lactate | pre-intervention and immediately after the intervention
  Lactate concentration (mmol/L) will be performed through blood extractions and measured using the YSI 2500

OTHER OUTCOMES:
PHYSICAL ACTIVITY | pre-intervention
  With INTERNATIONAL PHYSICAL ACTIVITY QUESTIONNAIRE (IPAQ). IPAQ allows the indirect calculation of METs performed by a patient weekly, understanding MET as the ratio of the work metabolic rate to the resting metabolic rate. One MET is defined as 1 kcal/kg/hour and is roughly equivalent to the energy cost of sitting quietly. This scale would have a minimum of 0 METs and no maximum. Higher values mean greater activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Rodrigo Martin-San Agustin, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cuerda Del Pino A, Martin-San Agustin R, Jose Laguna Sanz A, Diez JL, Palanca A, Rossetti P, Gumbau-Gimenez M, Ampudia-Blasco FJ, Bondia J. Accuracy of Two Continuous Glucose Monitoring Devices During Aerobic and High-Intensity Interval Training in Individuals with Type 1 Diabetes. Diabetes Technol Ther. 2024 Jun;26(6):411-419. doi: 10.1089/dia.2023.0535. PMID 38215205